CLINICAL TRIAL: NCT00000945
Title: A Pilot Study of the Effect of Cidofovir for the Treatment of Progressive Multifocal Leukoencephalopathy (PML) in Subjects With Acquired Immunodeficiency Syndrome (AIDS)
Brief Title: A Study to Evaluate the Use of Cidofovir (an Experimental Drug) for the Treatment of Progressive Multifocal Leukoencephalopathy (PML) in AIDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 363; 11327 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Leukoencephalopathy, Progressive Multifocal
Keywords: Leukoencephalopathy, Progressive Multifocal; Probenecid; HIV-1; Central Nervous System Diseases; Acquired Immunodeficiency Syndrome; DNA, Viral; cidofovir; Anti-HIV Agents; Neurologic Examination; Renal Agents
MeSH Terms: conditions — HIV Infections; Leukoencephalopathy, Progressive Multifocal; Central Nervous System Diseases; Acquired Immunodeficiency Syndrome | interventions — Cidofovir; Probenecid

INTERVENTIONS:
Drug: Cidofovir
Drug: Probenecid

SUMMARY:
The purpose of this study is to evaluate the safety, tolerance, and overall effectiveness of cidovir to treat PML in AIDS patients.

PML is an opportunistic infection (HIV-associated, due to weak immune system) caused by a virus that attacks the brain. Cidovir has been used effectively to treat cytomegalovirus (CMV) of the eye. Cidovir could be an effective treatment for PML as well.

DETAILED DESCRIPTION:
PML is a demyelinating disease of the brain's white matter, occurring when the JC virus infects the brain of patients infected with HIV-1. Cidofovir is known to be an effective treatment for cytomegalovirus of the eye and, in laboratory and animal testing, has also been shown to be effective against several other viruses. However, cidofovir is considered investigational as a treatment for PML.

In this multicenter, open-label study 24 patients receive cidofovir iv over 1 hr on days 0, 7, then every 2 wk for a total of 13 doses.

Oral probenecid is given 3h prior to and 2h and 8h following cidofovir administration. Nucleoside and non-nucleoside reverse transcriptors are withheld on days of probenecid administration. Protease inhibitors are continued during probenecid administration.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have had symptoms of PML for no more than 90 days before study entry, or have had abnormal neurological exams related to PML.
* Have negative tests for bacterial or fungal infections.
* Agree to practice abstinence or use effective methods of birth control during the study.
* Are at least 18 years old.
* Have a life expectancy of at least 6 months.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of uveitis.
* Are allergic to sulfa drugs or probenecid.
* Have had active opportunistic infections other than Kaposi's sarcoma within 30 days before study entry.
* Have sickle cell anemia or trait.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marra CM, Study Chair; Barker DE, Study Chair
Locations (19):
- United States (19):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Kentucky Lexington, Cincinnati, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Marra CM, Rajicic N, Barker DE, Cohen BA, Clifford D, Donovan Post MJ, Ruiz A, Bowen BC, Huang ML, Queen-Baker J, Andersen J, Kelly S, Shriver S; Adult AIDS Clinical Trials Group 363 Team. A pilot study of cidofovir for progressive multifocal leukoencephalopathy in AIDS. AIDS. 2002 Sep 6;16(13):1791-7. doi: 10.1097/00002030-200209060-00012. PMID 12218391